CLINICAL TRIAL: NCT06744725
Title: Dual-function Semirigid Thoracoscopy Versus Semirigid Thoracoscopy for the Diagnosis of Pleural Diseases: A Protocol for a Multicenter Open-label Randomized Controlled Trial
Brief Title: Dual-function Semirigid Thoracoscopy Versus Semirigid Thoracoscopy for the Diagnosis of Pleural Diseases: A Multicenter Open-label Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2024-UE-1
Record Dates: First submitted 2024-12-09; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Pleural Diseases
MeSH Terms: conditions — Pleural Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dual-function semirigid thoracoscopy (Experimental): Patients received pleural biopsy using dual-function semirigid thoracoscopy.
  Interventions: Device: Pleural biopsy using dual-function semirigid thoracoscopy
- Semirigid thoracoscopy (Experimental): Patients received pleural biopsy using semirigid thoracoscopy
  Interventions: Device: Pleural biopsy using semirigid thoracoscopy

INTERVENTIONS:
Device: Pleural biopsy using dual-function semirigid thoracoscopy — Patients will receive pleural biopsy using dual-function semirigid thoracoscopy.
  Arms: Dual-function semirigid thoracoscopy
Device: Pleural biopsy using semirigid thoracoscopy — Patients received pleural biopsy using semirigid thoracoscopy
  Arms: Semirigid thoracoscopy

SUMMARY:
We designed and developed a novel dual-function semirigid thoracoscope (UE FET-680; UE Corporation, Zhejiang, China) with a straight channel adapted to flexible and rigid forceps for pleural biopsy. Our preclinical trial has proven that the dual-function semirigid thoracoscope has larger and deeper sampling while retaining the entire thoracic accessibility and flexible bronchoscopic maneuvering habits of the semirigid thoracoscope. We designed this study to directly compare the diagnostic yield, quality of sampling, and safety between the dual-function semirigid thoracoscope and semirigid thoracoscope.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Unilateral pleural effusion of unclear etiology after a less invasive diagnosis
* Fully informed of the purpose and method of the study, agreed to participate in the study, and signed an informed consent form.

Exclusion Criteria:

* PaO2/FiO2 < 300
* Tendency for uncontrolled bleeding, unstable cardiovascular status, or severe heart failure
* A complete pleural symphysis, where it is not possible to create a pneumothorax
* Refractory cough
* Eastern Cooperative Oncology Group performance status 4
* Disagreements regarding study participation
* Participation in other studies within three months without withdrawal or termination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 6 Month
  The diagnostic yield in this study was defined as the proportion of all individuals undergoing the diagnostic procedure under evaluation in whom a specific diagnosis is established.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lee P, Colt HG. Rigid and semirigid pleuroscopy: the future is bright. Respirology. 2005 Sep;10(4):418-25. doi: 10.1111/j.1440-1843.2005.00737.x. PMID 16135163
- [Result] Rozman A, Camlek L, Marc-Malovrh M, Triller N, Kern I. Rigid versus semi-rigid thoracoscopy for the diagnosis of pleural disease: a randomized pilot study. Respirology. 2013 May;18(4):704-10. doi: 10.1111/resp.12066. PMID 23418922
- [Result] Agarwal R, Aggarwal AN, Gupta D. Diagnostic accuracy and safety of semirigid thoracoscopy in exudative pleural effusions: a meta-analysis. Chest. 2013 Dec;144(6):1857-1867. doi: 10.1378/chest.13-1187. PMID 23928984
- [Result] Collins TR, Sahn SA. Thoracocentesis. Clinical value, complications, technical problems, and patient experience. Chest. 1987 Jun;91(6):817-22. doi: 10.1378/chest.91.6.817. PMID 3581930
- [Result] Venekamp LN, Velkeniers B, Noppen M. Does 'idiopathic pleuritis' exist? Natural history of non-specific pleuritis diagnosed after thoracoscopy. Respiration. 2005 Jan-Feb;72(1):74-8. doi: 10.1159/000083404. PMID 15753638
- [Result] Bhatnagar R, Maskell N. The modern diagnosis and management of pleural effusions. BMJ. 2015 Sep 8;351:h4520. doi: 10.1136/bmj.h4520. No abstract available. PMID 26350935